CLINICAL TRIAL: NCT01215032
Title: Prospective Study of Metformin in Castration-Resistant Prostate Cancer
Brief Title: Metformin in Castration-Resistant Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: slow accrual, competing clinical trials
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Dana-Farber Cancer Institute (Other); Brigham and Women's Hospital (Other); Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Matthew R. Smith, MD, PhD, Professor of Medicine, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-244
Record Dates: First submitted 2010-10-04; First posted 2010-10-05 (Estimated); Results first posted 2017-02-27 (Actual); Last update posted 2017-05-15 (Actual); Status verified 2017-04

CONDITIONS: Prostate Cancer
Keywords: castration-resistant prostate cancer; insulin levels; metformin
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Metformin (Experimental): This is the only arm of this phase 2 open label study
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — Taken orally twice daily each 28-day cycle, for 12 cycles

SUMMARY:
Metformin is a medication that is prescribed for people with diabetes to help the body respond better to its own insulin and decrease sugar production by the liver. This helps control the body's blood sugar level and is approved by the Food and Drug Administration (FDA) for the treatment of diabetes. Participant's in this research study will already be receiving androgen deprivation therapy (ADT) for prostate cancer. ADT is considered standard of care for prostate cancer. Changes in the participant's metabolism, including changes in insulin and blood sugar levels, are often seen as a result of this type of hormone therapy. Some studies have shown a relationship between insulin and prostate cancer. These studies have suggested that insulin may signal tumor cells to grow. Other studies suggest that people receiving metformin treatment for diabetes may enjoy better outcomes from their prostate cancer then other similar patients who are not treated with metformin.

DETAILED DESCRIPTION:
* Each treatment cycle lasts 4 weeks (28 days). Participants will take metformin twice a day for all 28 days (except for the first 7 days of the first cycle when they will take it just once daily.)
* The following procedures will be done on Day 1 of treatment cycles 1, 2, 4, 7 and 10: medical history review, performance status, physical exam, blood tests.
* If the participant's first computed tomography (CT) or bone scan at the time of screening showed evidence of cancer, CT and bone scans will be repeated on Day 1 of treatment cycles 4, 7 and 10.
* Participants will be in this research study for about 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the prostate
* History of bilateral orchiectomies or ongoing treatment with a GnRH agonist for GnRH antagonist
* Disease progression according to PSA Working Group 2
* Minimum starting PSA (Prostate Specific Antigen) level of 2.0 ng/mL
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0 or 1

Exclusion Criteria:

* Symptomatic metastases
* Receiving any other agents for the treatment of prostate cancer except gonadotropin releasing hormone (GnRH) agonist or antagonist within the last 30 days
* Received any investigational cancer treatment agents within the last 30 days
* Prior treatment with docetaxel
* History of diabetes requiring drug therapy
* Current treatment with metformin or metformin treatment within the last year
* History of allergic reaction to metformin
* Have uncontrolled intercurrent illness including, but not limited to ongoing or unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Serum creatinine 1.5mg/dL or greater
* Hepatic impairment
* Need for ongoing treatment with cimetidine
* History of a different malignancy except for the following circumstances: Individuals with a history of other malignancies are eligible of they have been disease-free for at least 5 years and are deemed by the investigator to be at low risk for recurrence of that malignancy. Individuals with the following cancers are eligible if diagnosed and treated within the past 5 years: basal cell or squamous cell carcinoma of the skin

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2010-09; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew R. Smith, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Metformin: This is the only arm of this phase 2 open label study
  Metformin: Taken orally twice daily each 28-day cycle
Period: Overall Study
Arm/Group | Metformin
Started | 21
Completed | 1
Not Completed | 20
Not completed — Adverse Event | 3
Not completed — Lack of Efficacy | 17

BASELINE CHARACTERISTICS:
Arm/Group | Metformin
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.86 (7.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 18
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: PSA (Prostate Specific Antigen) Response
Description: Percent change in PSA from baseline to 12 weeks.
Time Frame: Approximately 12 weeks
Measure: Median (Full Range); unit: percentage of baseline PSA
Arm/Group | Metformin
Number analyzed (Participants) | 21
percentage of baseline PSA | 161 [96.1 to 309.5]

2. Secondary Outcome: Number of Participants With PSA Response
Description: PSA response is defined as a 50% decline from baseline confirmed by a second PSA value 4 weeks later.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Metformin
Number analyzed (Participants) | 21
Participants | 0

3. Secondary Outcome: Relationship Between Baseline Metabolomic Profile and PSA Response
Description: To determine the plasma metabolomic profiles associated with response to metformin using the Metabolon platform. The Metabolon platform is a proprietary technique of metabolic profiling using mass spectrometry coupled with liquid and/or gas chromatography and robust bioinformatics. The aim is to test the hypothesis that insulin level is a biomarker that predicts activity of metformin therapy for the treatment of castrate-resistant prostate cancer.
Time Frame: 2 years
Population: Data was not collected for this outcome measure because blood (plasma) samples were never run on the Metabolon platform, as the study was terminated early.
Arm/Group | Metformin
Number analyzed (Participants) | 0

4. Secondary Outcome: Percent Maintaining Glycemic Control
Description: To describe glycemic control as assessed by hemoglobin A1C. Glycemic control was defined as maintaining fasting plasma glucose levels less than or equal to 130 mg/dL. Plasma glucose levels were measured at baseline (prior to metformin dosing), pre-month 2, pre-month 4, pre-month 7, pre-month 10 and pre-month 13, and/or at off-study visit.
Time Frame: 2 years
Population: Participants were stratified based on baseline hemoglobin A1c. HbA1c < 6.0 is considered normal; HbA1c >/= 6.0 is considered abnormal.
Measure: Count of Participants; unit: Participants
Groups:
- Normal Baseline Hemoglobin A1c: Hemoglobin A1c less than 6.0 before metformin dosing began.
- Abnormal Baseline Hemoglobin A1c: Hemoglobin A1c greater than or equal to 6.0 before metformin dosing began.
Arm/Group | Normal Baseline Hemoglobin A1c | Abnormal Baseline Hemoglobin A1c
Number analyzed (Participants) | 15 | 6
Participants | 15 | 6

ADVERSE EVENTS:
Arm/Group | Metformin
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 16/21
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Metformin (N=21)
Hypothyroidism (Endocrine disorders) | 1
cataract (Eye disorders) | 1
abdominal pain (Gastrointestinal disorders) | 1
diarrhea (Gastrointestinal disorders) | 10
flatulence (Gastrointestinal disorders) | 2
frequent bowel movements (Gastrointestinal disorders) | 1
nausea (Gastrointestinal disorders) | 4
vomiting (Gastrointestinal disorders) | 1
chills (General disorders) | 1
fatigue (General disorders) | 4
fever (General disorders) | 1
Generalized achiness (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
anorexia (Metabolism and nutrition disorders) | 3
hyperglycemia (Metabolism and nutrition disorders) | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Buttock pain (Musculoskeletal and connective tissue disorders) | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Numbness in Toes (Musculoskeletal and connective tissue disorders) | 1
Numbness - buttocks (Musculoskeletal and connective tissue disorders) | 1
Urinary frequency (Renal and urinary disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
Early termination due to slow accrual led to small numbers of subjects. Therefore, meaningful assessment of the study endpoints is severely limited by the small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes